CLINICAL TRIAL: NCT03471195
Title: Salivary Cytokine Profile as Biomarker for Dental Pain in Children With Cerebral Palsy - An Exploratory Study
Brief Title: Salivary Cytokine Profile as a Biomarker for Dental Pain
Status: Completed | Type: Observational
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dr Sharat Pani, Program Director Pediatric Dentistry, Riyadh Colleges of Dentistry and Pharmacy
Other Study IDs: FPGRP/43635002/175
Record Dates: First submitted 2018-03-04; First posted 2018-03-20 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Cerebral Palsy; Dental Diseases
MeSH Terms: conditions — Cerebral Palsy; Stomatognathic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CP: A total of 20 children with cerebral palsy and dental decay will undergothe following Collection of Saliva Total Salivary Cytokine Profile
  Interventions: Diagnostic Test: Total Salivary Cytokine profile
- Control: A total of 20 verbal children without cerebral palsy matched for age and extent of dental decay will undergo the following Collection of Saliva Total Salivary Cytokine Profile
  Interventions: Diagnostic Test: Total Salivary Cytokine profile

INTERVENTIONS:
Diagnostic Test: Total Salivary Cytokine profile — Saliva will be collected using the passive drool technique and stored in a deep freezerat-60C.
  Other Names: cytokine profile

SUMMARY:
always reliable.Pain is an important diagnostic tool in dentistry. The type of treatment, extent of treatment and, sometimes, even the decision on whether to treat or not is dependent on the pain history obtained from the patient.The absence of an accurate description of dental pain is a factor that severely limits dental treatment planning in children with CP. The aim of this study is to study to evaluate the salivary cytokine profile of children with CP who have severe dental problems and to compare this to verbal children who have a similar dental profile.

DETAILED DESCRIPTION:
The sample with CP will be selected from individuals attending the dental clinics of the Prince Sultan bin Abdulaziz Humanitarian city (SBAHC). The control patients will be selected from the dental clinics of the Riyadh Colleges of Dentistry and Pharmacy and be matched to the CP patients for age, gender and extent of dental problems. The sample will comprise of 20 patients with CP and 20 verbal controls.The oral health of all children will be recorded using WHO examination criteria .The teeth will be examined using WHO category II criteria - clinical examination with lighting and without radiographs.aliva will be collected from the children using the passive drool method and stored in sterile plastics collection tubes. The collected sample will be stored at -600C until they can be analyzed. The cytokine profile of the saliva sample will be analyzed using an ELISA kit for total cytokine profile (Luminex Performance Human Cytokine Panel A, LUH000, R&D systems) to measure cytokines IL-1 alpha, IL-1 beta, IL-8, and TNF-alpha. The pain perception of the verbal control group will be recorded using the validated Arabic version of the short form of the McGill Pain Questionnaire. The children will also indicate the extent of the pain using the Wong Baker Faces ™ pain perception scale.Normality of the total cytokine levels will be tested using the Shapiro-Wilkes Test. The Mann Whiney U test will be used to compare the cytokine profile the CP and control group. The spearman correlation will be used to explore the relationship between the reported pain and cytokine profile levels. If found to be significant an initial cytokine-pain map will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* At least one tooth with pulpal involvement
* Aged between 8-12 years
* No neurological illness (for Control Group)
* Ability to verbalize pain (for Control Group)
* One dental tooth with pulpal involvement matching the condition of the test group (for Control Group)

Exclusion Criteria:

* confounding neurological disorders
* History of orofacial pain syndromes
* Absence of consent or assent

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will comprise of children with cerebral palsy(unable to verbalize pain) who have at least one dental condition that would be considered painful.
  The sample will be matched to controls who have similar dental status and can verablize pain
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Salivary Cytokine profile | 0 weeks (baseline)
  Salivary IL1alpha in mcg, Salivary IL1beta in mcg, Salivary IL6 in mcg, IL8 in mc , Salivary TNFalpha in mcg

CONTACTS AND LOCATIONS:
Overall Officials: Hezekiah A Mosadomi, DMD, Study Chair — Riyadh Elm University
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No